CLINICAL TRIAL: NCT00820235
Title: Prospective, Comparative Assessment of Single-tooth Replacement in Different Implant-abutment Settings
Brief Title: Study Comparing Appearance and Function of Three Different Dental Implant Designs When Placed in Front Region of Upper Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0003
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Device: OsseoSpeed™
- B (Active Comparator)
  Interventions: Device: NobelSpeedy™ Replace®
- C (Active Comparator)
  Interventions: Device: NanoTite™ Certain® PREVAIL®

INTERVENTIONS:
Device: OsseoSpeed™ — OsseoSpeed™ implant
  Arms: A
Device: NobelSpeedy™ Replace® — NobelSpeedy™ Replace® implant
  Arms: B
Device: NanoTite™ Certain® PREVAIL® — NanoTite™ Certain® PREVAIL® implant
  Arms: C

SUMMARY:
The primary objective is to compare the gum response to three different dental implant designs when placed in the front region of the upper jaw. The changes from baseline to one year after will be compared. The null-hypothesis is that the buccal soft tissue (gum) changes from baseline to one year after are equal for all three implant-abutment interface settings.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* At least 18 years
* In need of one or more single implants replacing missing or non-restorable teeth in the maxilla within region 14 to 24

The following should be considered at inclusion but can not be fulfilled until at Visit 2:

* Edentulous for at least 5 months at study site
* A buccal-lingual bone width at study site of at least 5.5 mm
* A mesial-distal bone level distance between adjacent teeth at study site of at least 5.5 mm
* A keratinized mid-buccal mucosal height of at least 2 mm at study site
* Teeth adjacent (mesial and distal) to study site must consist of two stable teeth on natural roots without signs of periodontal bone loss (>1 mm) and/or significant soft tissue loss
* Teeth adjacent (mesial and distal) to study site must demonstrate a stable occlusal guidance that will allow non-functional disclusion in all eccentric positions
* An opposing dentition with teeth, implants or prosthesis

Exclusion Criteria:

* Insufficient interocclusal distance for implant placement and restoration at study site
* Tooth adjacent (mesial and/or distal) to study site is ankylosed
* More than 2 mm vertical bone loss at study site as measured from the mid-buccal crest of bone on the adjacent teeth
* Site development (bone tissue) performed at less than 5 months before Visit 2 at study site
* Untreated rampant caries and/or uncontrolled periodontal disease
* Class II division 2 malocclusion (Edward Hartley Angle)
* Use of tobacco within last 6 months
* Uncontrolled diabetes (subjects history does not reveal the absence of control of insulin-dependent/non-insulin dependent Diabetes Mellitus)
* Current alcohol or drug abuse
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Use of any substance that will influence bone metabolism
* Need for systemic corticosteroids or any other medication that would influence post-operative healing and/or osseointegration
* History of radiation in the head and neck region
* Known pregnancy, pregnancy tests will be performed as per local requirements.
* Unable or unwilling to return for follow-up visits for a period of 5 years
* Unlikely to be able to comply with study procedures according to Investigators judgement
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study center)
* Previous enrollment or randomization of treatment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Cooper, Prof., Study Director — University of Illinois College of Dentistry
Locations (4):
- United States (3):
  - University of Iowa, College of Dentistry, Iowa City, Iowa
  - University of North Carolina, School of Dentistry, Chapel Hill, North Carolina
  - Perio Health Clinical Research Center, Houston, Texas
- Faculty of Dentistry, McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Result] McGuire MK, Scheyer T, Ho DK, Stanford CM, Feine JS, Cooper LF. Esthetic outcomes in relation to implant-abutment interface design following a standardized treatment protocol in a multicenter randomized controlled trial--a cohort of 12 cases at 1-year follow-up. Int J Periodontics Restorative Dent. 2015 Mar-Apr;35(2):149-59. doi: 10.11607/prd.2341. PMID 25738335
- [Result] Cooper LF, Reside G, Stanford C, Barwacz C, Feine J, Abi Nader S, Scheyer ET, McGuire M. A multicenter randomized comparative trial of implants with different abutment interfaces to replace anterior maxillary single teeth. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):622-32. doi: 10.11607/jomi.3772. PMID 26009913
- [Result] Barwacz CA, Stanford CM, Diehl UA, Qian F, Cooper LF, Feine J, McGuire M. Electronic assessment of peri-implant mucosal esthetics around three implant-abutment configurations: a randomized clinical trial. Clin Oral Implants Res. 2016 Jun;27(6):707-15. doi: 10.1111/clr.12640. Epub 2015 Jun 21. PMID 26096162

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- Group-A. OsseoSpeed™ Implant: Subjects that had OsseoSpeed™ implants installed.
- Group-B. NobelSpeedy™ Replace® Implant: Subjects that had NobelSpeedy™ Replace® implants installed
- Group-C. NanoTite™ Certain® PREVAIL® Implant: Subjects that had NanoTite™ Certain® PREVAIL® implants installed
Period: Overall Study
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Started | 48; 48 Implants | 49; 49 Implants | 44; 44 Implants
Completed | 33; 33 Implants | 28; 28 Implants | 27; 27 Implants
Not Completed | 15; 15 Implants | 21; 21 Implants | 17; 17 Implants

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant | Total
Number analyzed (Participants) | 48 | 49 | 44 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15) | 46 (17) | 46 (16) | 45 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 35 | 22 | 80
  Male | 25 | 14 | 22 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 5 | 10
  White | 42 | 46 | 36 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 9 | 7 | 26
  United States | 38 | 40 | 37 | 115

OUTCOME MEASURES:

1. Primary Outcome: Buccal Soft Tissue (Gum) Changes, Measured as Mid-buccal Gingival Zenith (GZ) Scores.
Description: Soft tissue response was evaluated by measuring it clinically and by evaluating it from clinical photographs using image analysis. Clinical evaluations of gingival zenith were performed at time of loading (permanent restoration) and at the 5-year follow-up after loading.
  The vertical distance from the most apical aspect of the soft tissue margin to the incisal edge of implant crown was measured using a standardized periodontal probe to the nearest half millimeter using the surgical loupe. The changes in the gingival zenith was calculated for each study position and the average for each treatment group was calculated for the evaluation period.
Time Frame: Evaluated at time of loading (permanent restoration) and at the 5-years follow-up after loading
Population: A total of 88 subjects completed the 5-year follow-up visit. Five radiographs (two in group A, two in group B and one in group C) were not possible to evaluate, giving an overall number of 83 subjects (83 implants) as basis for the analysis of Gingival Zenith score change.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Number analyzed (Participants) | 31 | 26 | 26
Number analyzed (Implants) | 31 | 26 | 26
Millimeter | 0.08 (0.65) | -0.10 (1.00) | 0.00 (0.58)

2. Secondary Outcome: Marginal Bone Level Alterations
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal Bone Level expressed in millimeters at the 5-year follow-up visit compared to values obtained at time of implant placement.
Time Frame: Evaluated at time of implant installation and at the 5-year follow-up visit.
Population: A total of 88 subjects completed the 5-year follow-up visit. Three radiographs (all in group C) were not possible to evaluate, giving an overall number of 85 subjects (85 implants) as basis for the analysis of marginal bone level change.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Number analyzed (Participants) | 33 | 28 | 24
Millimeter | -0.16 (0.45) | -0.92 (0.70) | -0.81 (1.06)

3. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of PPD
Description: Condition of the periimplant mucosa by assessment of probing pocket depth (PPD).
  Change in pocket depth expressed in millimeters at the 5-year follow-up visit, compared to values obtained at delivery of permanent restoration, i.e. loading (baseline).
  Negative value = increased pocket depth.
Time Frame: Measured at time of loading of permanent restoration and at the 5-year follow-up.
Population: A total of 88 subjects completed the 5-year follow-up visit. All those subjects are included in the PPD assessment.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Number analyzed (Participants) | 33 | 28 | 27
Millimeter | 0.08 (0.88) | -0.06 (0.88) | -0.09 (0.57)

4. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of Change in BoP.
Description: Condition of the periimplant mucosa by assessment of Bleeding on Probing (BoP). Presented as change in proportion of surfaces that show presence of BoP, measured from implant loading to the 5-year follow-up visit.
Time Frame: Measured at the implant loading and at the 5-year follow-up after loading.
Population: A total of 88 subjects completed the 5-year follow-up visit. All those subjects are included in the assessment of BoP change.
Measure: Mean (Standard Deviation); unit: Change in proportion of surfaces
Units Other Than Participants: Surfaces
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Number analyzed (Participants) | 33 | 28 | 27
Number analyzed (Surfaces) | 33 | 28 | 27
Change in proportion of surfaces | 0.13 (0.38) | 0.04 (0.34) | 0.07 (0.33)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group-A. OsseoSpeed™ Implant | Group-B. NobelSpeedy™ Replace® Implant | Group-C. NanoTite™ Certain® PREVAIL® Implant
Serious Adverse Events (participants affected / at risk) | 8/48 | 3/49 | 8/44
Other Adverse Events (participants affected / at risk) | 8/48 | 23/49 | 10/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A. OsseoSpeed™ Implant (N=48) | Group-B. NobelSpeedy™ Replace® Implant (N=49) | Group-C. NanoTite™ Certain® PREVAIL® Implant (N=44)
Breast cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalized due to fever after mastectomy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalized for partial nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalised for gall bladder surgery (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalized for follow-up on chest pains (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Hospitalized for spine fusion surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalized for gastric surgery (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalized for surgery of infected appendix (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalized for knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization after heart attack (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Death caused by heart attack (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalized due to episode of bi-polar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalized for fractured leg after an accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalized due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalized for treatment of infection after vaccination (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hospitalized due to menstrual hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A. OsseoSpeed™ Implant (N=48) | Group-B. NobelSpeedy™ Replace® Implant (N=49) | Group-C. NanoTite™ Certain® PREVAIL® Implant (N=44)
Study implant failled to osseointegrate (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 6 (6)
Study implant temporary mobile (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Restoration failure (Product Issues) | 6 (6) | 8 (8) | 1 (1) — Fractured/mobile/de-bonded dental crown on the study implant.
Loose abutments (Product Issues) | 3 (3) | 2 (2) | 0 (0) — Abutment screws temporarily loose
Other (General disorders) | 1 (1) | 9 (9) | 2 (2) — Mixed Adverse Events Pain (less the 5% per category). Including: swelling of soft tissue, bone loss around implant, fistula, infection, food impaction in tooth etc., etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less